CLINICAL TRIAL: NCT06168591
Title: Neuromuscular Impairment in Aging: a Longitudinal Study of Structural and Functional Mechanistic Bases of Age-related Alterations
Brief Title: Longitudinal Neuromuscular and Metabolic Changes With Aging
Acronym: TrajectorAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pavia (Other)
Collaborators: University of Padova (Other); Politecnico di Milano (Other); Turin, Italy (Other); University of Parma (Other)
Responsible Party: Principal Investigator, Simone Porcelli, Associate Professor, University of Pavia
Other Study IDs: UPavia-TrajectorAGE
Record Dates: First submitted 2023-11-24; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Aging; Muscle Physiology; Neurophysiology; Exercise Training; Sports Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ELDERLY: MIDDLE-AGED and OLD individuals of both sexes will be recruited. The stratification into ACTIVE and SEDENTARY will be done according to current public health guidelines

SUMMARY:
Ageing is characterized by a decline in neuromuscular control and a progressive loss of muscle mass, strength and power, leading to reduced mobility, loss of independence, higher hospitalizations rate, and increased all-cause mortality. Several studies suggest a non-linear decay of these age-related changes. Denervation-reinnervation processes, resulting in fewer but larger surviving motor units in advanced age, start as early as age 50-60yr and can be magnified in older adults (>75yr). Significant functional consequences in daily living activities are not usually observed until approximately 50yr. However, after 50yr, muscle strength/power reduction is accelerated and becomes faster than average muscle mass loss. Most observations come from cross- sectional studies and several confounding factors associated with secondary aging, such as physical activity levels, may contribute to (or compensate for) the observed age-related reductions in neuromuscular function. Compared to cross-sectional designs, prospective ones are advantageous in their ability to investigate fundamental mechanisms by excluding inter-subjects variability. In this project, the investigators will characterize longitudinal age-related changes in motor function, physical performance and muscle aerobic metabolism with an integrated approach. The investigators aim to combine classical methods of in-vivo and ex-vivo evaluation of neuromuscular function with innovative approaches for assessing changes and interactions between neural, structural and metabolic variables in two critical phases of ageing: 55-60yrs and 75-80yrs. Within each age-group, subjects will be classified based on their functional capabilities and divided in either active or sedentary. The investigators will describe the 2-yr time course of 1) mechanisms impairing neuromuscular function (denervation-reinnervation processes); 2) interactions between muscle structural changes and neural/metabolic impairments; 3) functional and metabolic changes occurring at whole muscle as well as single fibers level. The results will extend current understanding of physiological determinants of neuromuscular alterations in aging by identifying the course and rate of changes of specific factors that mediate functional loss and disability in older adults.

DETAILED DESCRIPTION:
State of the art The life expectancy of humans has continuously increased in most countries over the last century. With extended life expectancy, quality of life of elderly is a priority. However, ageing is a physiological process characterized by a decline in neuromuscular control and a progressive loss of muscle mass, strength and power. These impairments negatively affect mobility, increase morbidity and have dramatic individual and societal impacts.

On average, elderly walk more slowly, have less muscle strength and power, have poorer memory and reasoning abilities, and are slower to respond on speeded cognitive tasks relative to younger adults. In cross-sectional reports age-related changes in physical capability and associations between lower physical capability levels and higher mortality rates are consistently found. Nevertheless, there is a growing body of literature suggesting that chronological age alone cannot account for the heterogeneity in structural, functional, and physiological changes associated with human ageing.

One of the main neurophysiological mechanisms underlying the age-related changes in muscle function is the progressive loss of motor neurons, usually accompanied by instability of NMJ. The extent to which this phenomenon affects muscle structure, neuromuscular control and their interaction at different ageing phases is only partly described, also due to the wide inter-subject variability.

Moreover, in aged adults slower gait speed, lower muscle strength and changes in muscle quality have been correlated to impaired skeletal muscle oxidative capacity, with elderly showing lower O2 consumption at peak exercise and impaired submaximal muscle oxidative function compared to young.

The literature reports are mainly cross-sectional and factors associated with secondary aging such as physical activity levels may influence cross-sectional data. Thus, a longitudinal monitoring of neuromuscular and metabolic impairments in aging is needed, aiming to:

AIM 1 - Describe longitudinal age-related changes in motor function and physical performance with combined muscle mass and muscle aerobic metabolism AIM 2 - Identify the underlying mechanisms impairing in-vivo neuromuscular function by changes in muscle denervation and reinnervation AIM 3 - Define the role of skeletal muscle structural remodeling and muscle bioenergetics decline at whole-body level on neuromuscular impairments AIM 4 - Quantify functional and metabolic changes occurring at single muscle fibers level AIM 5 - Determine level of physical activity and related beneficial effects

ELIGIBILITY:
Inclusion Criteria:

Community dwelling, mobility and cognitively unimpaired participants will be enrolled. Cognitive assessment: Mini Mental Status Examination (MMSE, cutoff: 24). Physical performance assessments: gait speed over 4-m (WS, >0,8 m/s), Short Physical Performance Battery (SPPB, >9), the Timed-Up and Go test (TUG <20) and grip strength (GRIP, >27 kg (M) or >16 kg (F)).

Exclusion Criteria:

Parkinson's disease or other neurological disorder; diabetes; stroke; late-stage cancer; chronic kidney disease (IV and V stages); severe liver insufficiency; severe cardiac disorder and major recent heart surgery; severe osteoarthritis.

Ages: 55 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: MIDDLE-AGED (55-60yrs) and OLD (75-80yrs) individuals of both sexes will be recruited. The stratification into ACTIVE and SEDENTARY will be done according to current public health guidelines and accelerometric data.
  Participants will be recruited among subjects who routinely visit the facilities of the Clinical Unit of Geriatric for routine evaluations. If inclusion and exclusion criteria are matched, the level of physical activity will be monitored across 7 consecutive days by accelerometers and participants classified as SEDENTARY or ACTIVE.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Perceived quality of life by EQ-5D-5L | up to 24 months
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/ depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Muscle weakness Muscle strength | up to 24 months
  Muscle force production during isometric contraction
Exercise tolerance | up to 24 months
  Maximal oxygen consumption
Motor unit recruitment | up to 24 months
  Neuromuscular adaptations will be assessed using surface EMG detected with grids of electrodes
Muscle Architecture | up to 24 months
  Structural adaptations will be assessed in-vivo using Ultrasonography (US)

SECONDARY OUTCOMES:
Muscle oxidative capacity | up to 24 months
  Mitochondrial function will be estimated in vivo by near infrared spectroscopy
Physical activity behavior | up to 24 months
  Levels of physical activity will be monitor by accelerometric wearable devices
Endothelial function | up to 24 months
  Blood flow changes during leg passive movement will be recorded by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Lauretani, MD, Study Director — University of Parma
Locations (1):
- University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No